CLINICAL TRIAL: NCT04838639
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Food Effect of NO-13065 When Administered Orally to Healthy and Obese Adult Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Food Effect of NO-13065 in Healthy and Obese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Factory, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 360-101
Record Dates: First submitted 2021-03-30; First posted 2021-04-09 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2022-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NO-13065, oral tablet (Experimental)
  Interventions: Drug: NO-13065
- Placebo matched to NO-13065, oral tablet (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NO-13065 — Single ascending doses of NO-13065 in separate cohorts of subjects; each cohort consists of 6 subjects treated with NO-13065.
  Single ascending dose of NO-13065 with food effect arm. Multiple ascending doses of NO-13065 for 10 or up to 28 days in separate cohorts of subjects; each cohort consists of 6 subjects treated with NO-13065.
  Arms: NO-13065, oral tablet
Drug: Placebo — Two subjects per cohort will take a matched placebo.
  Arms: Placebo matched to NO-13065, oral tablet

SUMMARY:
This clinical trial is the first-in-human study of NO-13065. The purpose of this phase 1 study is to assess the safety and tolerability of single and multiple ascending oral doses and food effect of NO-13065 in healthy and obese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and/or female (non-childbearing potential only), 19 to 55 years of age
2. Continuous non-smoker
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or safety ECGs.
4. Women of non-childbearing potential only
5. Able to understand and sign a written informed consent form prior to initiation of study procedures.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems
2. History or presence of clinically significant medical or psychiatric condition or disease
3. History or presence : Familial hyperlipidemia, Diabetes, Bleeding disorder(s), including relevant familial history, Thromboembolic disease, Bleeding in the gastrointestinal tract or CNS, Hepatobillary disease, Gilbert's syndrome
4. History or presence of alcohol or drug abuse.
5. Has liver function test(s) including ALT, AST, GGT, and/or ALP or total bilirubin that are > ULN at screening or check-in.
6. Positive urine drug or alcohol results.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | Up to 35 days
  To assess the safety and tolerability of single and multiple ascending oral doses of NO-13065 in healthy, overweight, and obese adult subjects.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 35 days
  To assess Cmax of single and multiple ascending oral doses of NO-13065 in healthy, overweight, and obese adult subjects.
Area under the plasma concentration-time curve (AUC) | Up to 35 days
  To assess AUC of single and multiple ascending oral doses of NO-13065 in healthy, overweight, and obese adult subjects.
Time to reach Cmax (Tmax) | Up to 35 days
  To assess Tmax of single and multiple ascending oral doses of NO-13065 in healthy, overweight, and obese adult subjects.
Apparent first-order terminal elimination half-life (t ½) | Up to 35 days
  To assess t ½ of single and multiple ascending oral doses of NO-13065 in healthy, overweight, and obese adult subjects.
Correlation between QTc and NO-13065 plasma concentrations | Up to 29 days
  To explore the correlation between changes in QTc interval (msec) and NO-13065 plasma concentrations, appropriate correction method for QTc interval calculation such as QTcF will used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Koushi Iwata, Study Chair — Otsuka Pharmaceutical Factory, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No